CLINICAL TRIAL: NCT01741155
Title: A 2-Part Phase 2 Study of SPI-1620 in Combination With Docetaxel Versus Docetaxel Alone for Patients With Non Small-cell Lung Cancer After Failure of First-line Platinum-based Chemotherapy
Brief Title: Study of SPI-1620 in Combination With Docetaxel Versus Docetaxel Alone for Patients With Non Small-cell Lung Cancer (NSCLC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study did not meet efficacy end point and did not enroll patients in the randomized phase.
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPI-1620-12-201
Record Dates: First submitted 2012-11-27; First posted 2012-12-04 (Estimated); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Non Small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — sovateltide; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Single Arm Part: SPI-1620 & Docetaxel (Experimental): Patients will receive 11 μg/m2 of SPI-1620 IV followed by docetaxel 75 mg/m2 IV. Cycles will continue every 3 weeks until progression or intolerable toxicity.
  Interventions: Drug: SPI-1620; Drug: Docetaxel
- Randomized Part: SPI-1620 & Docetaxel (Experimental): Patients will receive 11 μg/m^2 of SPI-1620 intravenous (IV) followed by docetaxel 75 mg/m^2 IV administered in 3-week cycles until progression or intolerable toxicity.
  Interventions: Drug: SPI-1620; Drug: Docetaxel
- Randomized Part: Docetaxel (Active Comparator): Patients will receive 75 mg/m^2 docetaxel in 3-week cycles until progression or intolerable toxicity.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: SPI-1620 — SPI-1620 11 μg/m2 administered intravenously over one minute.
  Arms: Randomized Part: SPI-1620 & Docetaxel; Single Arm Part: SPI-1620 & Docetaxel
Drug: Docetaxel — Docetaxel: 75 mg/m2 administered as IV infusion.
  Other Names: Taxotere

SUMMARY:
The purpose of this study is to estimate and compare the objective response rate of SPI-1620 administered in combination with docetaxel in patients with NSCLC and to determine the safety of SPI-1620 when administered in combination with docetaxel.

DETAILED DESCRIPTION:
This will be a two part study. In Single Arm Part, patients will receive 11 μg/m2 of SPI-1620 IV followed by docetaxel 75 mg/m2 IV. Cycles will continue every 3 weeks until progression or intolerable toxicity. Overall 27 patients will be enrolled in the Single Arm Part. If 6 or more responses (CR/PR) are observed in this group then the Randomized Part will be initiated.

In the Randomized Part approximately 200 patients (100 per arm) will be randomized to receive SPI-1620 plus docetaxel or docetaxel alone.

In the experimental arm, patients will receive 11 μg/m2 of SPI-1620 IV followed by docetaxel 75 mg/m2 IV administered in 3-week cycles until progression or intolerable toxicity. In the control arm, patients will receive 75 mg/m2 docetaxel in 3-week cycles until progression or intolerable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed locally advanced or metastatic NSCLC that has failed one prior platinum-containing chemotherapy
* Measurable disease as per RECIST v. 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
* Adequate bone marrow, liver and renal function

Exclusion Criteria:

* More than one prior chemotherapy regimen for metastatic NSCLC
* Known, uncontrolled central nervous system (CNS) metastases
* Significant circulatory disorders in the past 6 mo.
* Concomitant treatment with phosphodiesterase inhibitors
* Uncontrolled orthostatic hypotension, asthma or chronic obstructive pulmonary disease (COPD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) of SPI-1620 | Up to 2 years
  To estimate and compare the objective response rate of SPI-1620 administered in combination with docetaxel in patients with NSCLC

SECONDARY OUTCOMES:
Duration of Response (DoR) | Up to 12 weeks
  only in Randomized Part.
Progression-free survival(PFS) | 2 years from the start of study treatment
  only in Randomized Part
Overall survival (OS) | 2 years from the start of study treatment
Safety of SPI-1620 | Up to 2 years
  Periodic physical examinations with vital sign monitoring, safety laboratories and monitoring of adverse events will be performed.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Oncology Hematology Care Inc., Cincinnati, Ohio
  - Tennessee Oncology PLLC, Chattanooga, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - Virginia Cancer Institute, Richmond, Virginia